CLINICAL TRIAL: NCT01211002
Title: The Exploratory Clinical Study of Concurrent Chemo-radiotherapy Combined With Recombinant Human Endostatin (Endostar) for Local Advanced Non-small Cell Lung Cancer (NSCLC (Ⅲ A / Ⅲ B) )
Brief Title: Study of Concurrent Chemo-radiotherapy Combined With Recombinant Human Endostatin for Local Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Simcere Pharmaceutical Co., Ltd (Other)
Collaborators: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Zhenzhou Yang M.D., Daping Hospital and Research Institute of Surgery of Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sim201002
Record Dates: First submitted 2010-09-27; First posted 2010-09-29 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Radiotherapy; rh-endostatin; chemotherapy; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy; Endostatins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- radiotherapy combined with EP (Active Comparator): the dose of radiotherapy is 60-66 Gy / 30-33f.The combination regimen is etoposide (50 mg/m2 day1-5, 29-33) and cisplatin (50 mg/m2 day1, 8, 29, 36) in the 1st, 4th weeks of radiotherapy for 2 courses.
  Interventions: Radiation: radiotherapy combined with EP
- adiotherapy / EP /recombinant human endostatin (Experimental): recombinant human endostatin: The number of courses is 3 ~ 4 and each course last for 28 days.dose:15mg，d1-14, intravenous injection.
  Interventions: Drug: radiotherapy / EP combined with recombinant human endostatin

INTERVENTIONS:
Radiation: radiotherapy combined with EP — Tumor vo lume is 60-66 Gy / 30-33f and the combination regimen is etoposide (50 mg/m2 day1-5, 29-33) and cisplatin (50 mg/m2 day1, 8, 29, 36) in the 1st, 4th weeks of radiotherapy for 2 courses.
  Arms: radiotherapy combined with EP
Drug: radiotherapy / EP combined with recombinant human endostatin — Anti-vascular targeting therapy The number of courses is 3 ~ 4 and each course last for 28 days. Recombinant human endostatin（Endostar）：15mg，d1-14, intravenous injection.
  Arms: adiotherapy / EP /recombinant human endostatin

SUMMARY:
It is a trials to evaluate the overall survival (OS) of radiotherapy / EP combined with recombinant human endostatin in treatment of locally advanced (Ⅲ A / unresectable Ⅲ B) non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically or histologically confirmed and inoperable stage Ⅲ (Ⅲ A or unresectable Ⅲ B) NSCLC;
2. Patients with ages of 18~70 years, general condition ECOG performance scale （PS）≤ 1, weight loss <10% during last 6 months;
3. CT films of patients during last 4 weeks were accessible when patients were selected into the groups, the lesions were measurable; (According to the standard of RECIST1.1, they should have at least one of accurately measurable lesions with the largest diameter ≥ 10mm by spiral CT, PET-CT, with the largest diameter≥ 20mm by ordinary CT and MRI.）
4. No major organ dysfunction, the function of heart, liver and kidney was normal, laboratory indicators should meet the following requirements: Blood: WBC> 4.0 × 109 / L, absolute neutrophil count > 1.5 × 109 / L, platelet count> 100 × 109 / L, hemoglobin> 110g / L; liver function: serum bilirubin was less than 1.5 × maximum normal value ; ALT and AST were less than 1.5 × maximum normal value; BUN, Cr within the normal range; FEV1 > 1L or> 40% of predicted value;
5. Patients could understand the circumstances of this study and those who have signed the informed consent form;

Exclusion Criteria:

1. Pregnant or lactating women; women of child-bearing age without contraception;
2. Acute infection or other serious underlying diseases;
3. Significant neurological, psychiatric history, including dementia which may influence the ability to understand and the informed consent;
4. Receive the treatment of other experimental trials in the same period; on the medication of other anticancer drugs a the same time; have joined other drug clinical trials 30 days before this clinical trial;
5. Diabetes without control (blood-glucose is unstable or ≥ 8mol / L after administration);
6. Patients who are allergic to E. coli preparation;
7. Patients who are unsuitable to participate in this trial determined by the researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | 3 years

SECONDARY OUTCOMES:
quality of life | 2 years
objective response rate (ORR) | 1 years
disease control rate (DCR) | 1 year
progression-free survival (PFS) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: zhenzhou yang, M.D., Study Chair — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Daping Hospital, Chongqin, China